CLINICAL TRIAL: NCT03539718
Title: Taurolidine Citrate and Unfractionated Heparin Combination Versus Unfractionated Heparin Alone in Prevention of Inflammation in Hemodialysis Catheters.
Brief Title: Taurolock Hep 500 Versus Unfractionated Heparin as Anti-inflammatory in Hemodialysis Catheters.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, amr mohamed mansour, Assistant Lecturer of nephrology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: taurolock hep 500 efficacy
Record Dates: First submitted 2017-07-31; First posted 2018-05-29 (Actual); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Hemodialysis Catheter Infection; Thrombosis; Dialysis Catheter
MeSH Terms: conditions — Thrombosis | interventions — Heparin

STUDY DESIGN:
Intervention Model Description: comparative
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- cases (Experimental): Cases, taurolidine heparin 500 will be used at end of session
  Interventions: Drug: Taurolidine heparin
- control (Active Comparator): Controls, Heparin Sodium 5000 will be given at end of session
  Interventions: Drug: Heparin Sodium

INTERVENTIONS:
Drug: Taurolidine heparin — Taurolock-hep 500 at end of session
  Other Names: Tautolock HEP 500
  Arms: cases
Drug: Heparin Sodium — Heparin sodium 5000 at end of session
  Other Names: Heparin Sodium 5000
  Arms: control

SUMMARY:
To assess the efficacy of Taurolock-hep500™ as anticoagulant and antimicrobial catheter lock solution in comparison to unfractionated heparin as alock solution to improve performance of hemodialysis catheters and quality of hemodialysis .

DETAILED DESCRIPTION:
In this study,investigators will recruit 60 patients with ESRD on regular hemodialysis from hemodialysis units in Ain-Shams university Hospitals, Patients will be recruited to study at the time of catheter insertion.

They will be randomized into 2 groups. Group 1; 30 Patients will receive unfractionated heparin (5000i.u/ml) after hemodialysis sessions (control group).

Group 2; 30 Patients will receive Taurolock-hep500™ after hemodialysis sessions. All patients will be subjected to;

1. Full history including history of ESRD and dialysis initiation.
2. Clinical examination. Aseptic technique will be used in handling with catheters including (sterile gloves, antiseptic solution in dealing with covers and caps topical antibiotics spray and ointment) catheter will be instilled by 10 ml of normal saline in both opening followed by either taurolock hep 500™ or unfractionated heparin 5000 iu/ml.

Patients will be followed up for one month and will be monitored for clinical symptoms and signs of catheter related bacteremia (fever ,rigors, hypotension, sweating ) on the hemodialysis sessions . Also catheter performance will be assessed using the following parameters;

1. Blood flow rate measured by hemodialysis machine blood pump in (ml/min).
2. Dialysis quality by URR( urea reduction ratio) is a dimensionless number used to quantify dialysis treatment adequacy by calculating difference between urea level before and after hemodialysis session (average of 4 sessions , 1 per each week).
3. CBC ,markers of inflammation (CRP) baseline and at time of appearance of symptoms and signs of bacteremia in both groups in addition to (IL6) measured by Elisa technique baseline and at time of appearance of symptoms and signs .

ELIGIBILITY:
Inclusion Criteria:

1. Patients on regular hemodialysis 3sessions/wk.
2. Recent catheter insertion at beginning of the study.
3. Both males and females.
4. Age group ≥ 18 ys.

Exclusion Criteria:

1. Patients with intercurrent infections.
2. Patients with sepsis.
3. Patients receiving drugs affecting immune system like immunosuppressive drugs.
4. Patients on antibiotics.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-05-15 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Prevention of inflammation in hemodialysis patients through hemodialysis catheters | one month
  Comparing levels of highly sensitive c-reactive protein and interleukin-6 levels before and after using the drug Urea reduction ratio over sessions

CONTACTS AND LOCATIONS:
Overall Officials: Magdy Sharkawy, MD, Study Director — Ain Shams University
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] FOGARTY, DAMIAN, and PETER MAXWELL.